CLINICAL TRIAL: NCT00528580
Title: Statins for the Early Treatment of Sepsis
Acronym: SETS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15420A
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Results first posted 2018-06-07 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Sepsis
Keywords: Sepsis; Statin; Infection; Immunomodulatory
MeSH Terms: conditions — Sepsis; Infections | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 (Experimental): Simvastatin 80 mg once daily PO (or via NG or G-tube)
  Interventions: Drug: Simvastatin
- 2 (Placebo Comparator): Identical-appearing placebo PO (or via NG or G-tube)
  Interventions: Drug: Identical-appearing placebo

INTERVENTIONS:
Drug: Simvastatin — 80 mg once daily PO/NG x 4 days
  Arms: 1
Drug: Identical-appearing placebo — once daily x 4 days
  Arms: 2

SUMMARY:
We propose a Phase II, randomized, placebo-controlled clinical trial to test the hypothesis that treatment with once-daily statins has a beneficial effect on inflammatory cytokines and clinical outcomes in adults hospitalized with sepsis. As our animal models suggest pretreatment with statins are required for their beneficial effects, we propose a study design intended to identify patients and initiate treatment early in their hospital stay. This Phase II study is intended to assess the feasibility of conducting a large-scale investigator-initiated translational research protocol that involves multiple clinical services within the Department of Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Initial presentation to the Emergency Department or University of Chicago MD office/Dialysis Center for current hospital admission
* Sepsis (ACCP/SCCM criteria)

  1. Clinically suspected infection as per the treating physician or confirmed infection
  2. 2 or more of the following: Temperature 38ºC (100.4ºF)or 36ºC (96.8ºF), Heart rate (HR) > 90/min, Respiratory rate (RR) > 20/min or PaCO2 < 32 mmHg, White blood cell count > 12,000/mm3 or < 4000/m3 or > 10%immature neutrophils
* Initiation of antibiotics by treating physician for sepsis
* Hospitalized from the Emergency Department or University of Chicago MD office/Dialysis Center to an inpatient medical service (intensive care unit (ICU)or non-ICU service) OR admission to the medical ICU (MICU) from a non-ICU inpatient medical floor.
* Assent of the primary treating physician at the time of enrollment.
* The meeting of SIRS criteria is due to an infection as per the treating physician.

Exclusion Criteria:

* Pregnancy
* ALT >3 times above the upper limit of normal
* Elevated creatine phosphokinase (CPK) (>3 times the upper limit of normal)
* Concurrent treatment with any of the following drugs: daptomycin, fenofibrate, ketoconazole,triaconazole, amiodarone, clarithromycin, cyclosporine, erythromycin,nefazodone, niacin, protease inhibitors, telithromycin, verapamil,danazol, gemfibrozil
* History of allergy or intolerance to statins
* Greater than 16 hours after meeting inclusion criteria
* Use of 1 more doses of statins in the previous 4 weeks
* Clinical indication for treatment with statin during hospital admission (per treating physician)
* Sufficiently poor prognosis prior to enrollment that treating physicians have elected to employ comfort care or plan to discharge to hospice
* Transfer from surgical service to medical service
* Needing transfusion for either active bleeding or severe hemolysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Krishnan, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Oba Y, Salzman GA. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury. N Engl J Med. 2000 Sep 14;343(11):813; author reply 813-4. No abstract available. PMID 10991706
- [Background] Almog Y, Shefer A, Novack V, Maimon N, Barski L, Eizinger M, Friger M, Zeller L, Danon A. Prior statin therapy is associated with a decreased rate of severe sepsis. Circulation. 2004 Aug 17;110(7):880-5. doi: 10.1161/01.CIR.0000138932.17956.F1. Epub 2004 Aug 2. PMID 15289367
- [Background] American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference: definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. Crit Care Med. 1992 Jun;20(6):864-74. PMID 1597042
- [Background] Dunbar LM, Wunderink RG, Habib MP, Smith LG, Tennenberg AM, Khashab MM, Wiesinger BA, Xiang JX, Zadeikis N, Kahn JB. High-dose, short-course levofloxacin for community-acquired pneumonia: a new treatment paradigm. Clin Infect Dis. 2003 Sep 15;37(6):752-60. doi: 10.1086/377539. Epub 2003 Aug 28. PMID 12955634
- [Background] Greenwood J, Walters CE, Pryce G, Kanuga N, Beraud E, Baker D, Adamson P. Lovastatin inhibits brain endothelial cell Rho-mediated lymphocyte migration and attenuates experimental autoimmune encephalomyelitis. FASEB J. 2003 May;17(8):905-7. doi: 10.1096/fj.02-1014fje. Epub 2003 Mar 5. PMID 12626426
- [Background] Gupta R, Plantinga LC, Fink NE, Melamed ML, Coresh J, Fox CS, Levin NW, Powe NR. Statin use and sepsis events [corrected] in patients with chronic kidney disease. JAMA. 2007 Apr 4;297(13):1455-64. doi: 10.1001/jama.297.13.1455. PMID 17405971
- [Background] Hackam DG, Mamdani M, Li P, Redelmeier DA. Statins and sepsis in patients with cardiovascular disease: a population-based cohort analysis. Lancet. 2006 Feb 4;367(9508):413-8. doi: 10.1016/S0140-6736(06)68041-0. PMID 16458766
- [Background] Jacobson JR, Barnard JW, Grigoryev DN, Ma SF, Tuder RM, Garcia JG. Simvastatin attenuates vascular leak and inflammation in murine inflammatory lung injury. Am J Physiol Lung Cell Mol Physiol. 2005 Jun;288(6):L1026-32. doi: 10.1152/ajplung.00354.2004. Epub 2005 Jan 21. PMID 15665042
- [Background] Leung BP, Sattar N, Crilly A, Prach M, McCarey DW, Payne H, Madhok R, Campbell C, Gracie JA, Liew FY, McInnes IB. A novel anti-inflammatory role for simvastatin in inflammatory arthritis. J Immunol. 2003 Feb 1;170(3):1524-30. doi: 10.4049/jimmunol.170.3.1524. PMID 12538717
- [Background] Liappis AP, Kan VL, Rochester CG, Simon GL. The effect of statins on mortality in patients with bacteremia. Clin Infect Dis. 2001 Oct 15;33(8):1352-7. doi: 10.1086/323334. Epub 2001 Sep 20. PMID 11565076
- [Background] Majumdar SR, McAlister FA, Eurich DT, Padwal RS, Marrie TJ. Statins and outcomes in patients admitted to hospital with community acquired pneumonia: population based prospective cohort study. BMJ. 2006 Nov 11;333(7576):999. doi: 10.1136/bmj.38992.565972.7C. Epub 2006 Oct 23. PMID 17060337
- [Background] Merx MW, Liehn EA, Graf J, van de Sandt A, Schaltenbrand M, Schrader J, Hanrath P, Weber C. Statin treatment after onset of sepsis in a murine model improves survival. Circulation. 2005 Jul 5;112(1):117-24. doi: 10.1161/CIRCULATIONAHA.104.502195. PMID 15998696
- [Background] Naidu BV, Woolley SM, Farivar AS, Thomas R, Fraga C, Mulligan MS. Simvastatin ameliorates injury in an experimental model of lung ischemia-reperfusion. J Thorac Cardiovasc Surg. 2003 Aug;126(2):482-9. doi: 10.1016/s0022-5223(03)00699-8. PMID 12928648
- [Background] Schmidt H, Hennen R, Keller A, Russ M, Muller-Werdan U, Werdan K, Buerke M. Association of statin therapy and increased survival in patients with multiple organ dysfunction syndrome. Intensive Care Med. 2006 Aug;32(8):1248-51. doi: 10.1007/s00134-006-0246-y. Epub 2006 Jun 21. PMID 16788803
- [Background] Thomsen RW, Hundborg HH, Johnsen SP, Pedersen L, Sorensen HT, Schonheyder HC, Lervang HH. Statin use and mortality within 180 days after bacteremia: a population-based cohort study. Crit Care Med. 2006 Apr;34(4):1080-6. doi: 10.1097/01.CCM.0000207345.92928.E4. PMID 16484926
- [Background] Yasuda H, Yuen PS, Hu X, Zhou H, Star RA. Simvastatin improves sepsis-induced mortality and acute kidney injury via renal vascular effects. Kidney Int. 2006 May;69(9):1535-42. doi: 10.1038/sj.ki.5000300. PMID 16557230
- [Derived] Dobesh PP, Olsen KM. Statins role in the prevention and treatment of sepsis. Pharmacol Res. 2014 Oct;88:31-40. doi: 10.1016/j.phrs.2014.04.010. Epub 2014 May 2. PMID 24794878

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled 2008-2009 at University of Chicago and Mercy Hosptial in Chicago, IL
Groups:
- Experimental: Simvastatin 80 mg once daily PO (or via NG or G-tube)
  Simvastatin: 80 mg once daily PO/NG x 4 days
- Placebo: Identical-appearing placebo PO (or via NG or G-tube)
  Identical-appearing placebo: once daily x 4 days
Period: Overall Study
Arm/Group | Experimental | Placebo
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Placebo | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 34 | 68
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (8) | 52 (8) | 52 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 17 | 17 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Time to Clinical Stability
Description: Normalization of vital signs for each subject enrolled. This is expressed as a mean time to normalization for each +/- standard error.
Time Frame: 24 hours
Measure: Mean (Standard Error); unit: days
Groups:
- Treatment Group: Simvastatin 80 mg once daily PO (or via NG or G-tube)
  Simvastatin: 80 mg once daily PO/NG x 4 days
- Control Group: Identical-appearing placebo PO (or via NG or G-tube)
  Identical-appearing placebo: once daily x 4 days
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 34 | 34
days | 3 (1) | 3 (1)

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Simvastatin: Simvastatin 80 mg once daily PO (or via NG or G-tube)
  Simvastatin: 80 mg once daily PO/NG x 4 days
Arm/Group | Simvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes